CLINICAL TRIAL: NCT01011023
Title: Unnecessary Gastric Decompression in Distal Elective Bowel Anastomoses in Children. A Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: DAVILA-PEREZ ROBERTO, PEDIATRIC SURGERY DEPARTMENT HOSPITAL INFANTIL DE MEXICO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: robdape1
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Unnecessary Nasogastric Tube; Bowel Anastomosis
Keywords: Bowel anastomosis; nasogastric tube; children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WITHOUT NASOGASTRIC TUBE (Experimental): 1. Experimental group (EG): without NGT, by removing the NGT at the end of the surgery, once the stomach had been aspirated,
  Interventions: Other: Non application of nasogastric tube in the experimental group
- WITH NASOGASTRIC TUBE (Active Comparator): 2. Control group (CG): with NGT, with radiographic corroboration of correct placement after the surgery. Both groups were given: 5-day fasting because it was the therapeutic gold standard at our hospital and our country, intravenous solutions and antibiotics for 5 days, ranitidine, and analgesics, without use of any antiemetic drug. Once the fasting period ended, in the CG the NGT was clamped and withdrawn, and in both groups oral fluids and diet were started. Once the regular diet was tolerated, the patients were discharged and followed up at clinic 30 days afterwards.
  Interventions: Other: Non application of nasogastric tube in the experimental group

INTERVENTIONS:
Other: Non application of nasogastric tube in the experimental group — Avoid the 5 post operative application of nasogastric tube in the experimental group vs the control group with the usual nasogastric tube

SUMMARY:
Objective. To study the role of nasogastric drainage to prevent postoperative complications in children with <b>distal</b> elective bowel anastomosis. Summary Background Data. Nasogastric drainage has been used as a routine measure after gastrointestinal surgery in children and adults, to hasten bowel function, prevent post operative complications and shorten hospital stay. However, there is no former study that states in a scientific manner its benefit in children. Methods. The investigators performed a clinical controlled, randomized trial, comprising 60 children that underwent distal elective bowel anastomoses comparing post operative complications between a group with nasogastric tube in place (n=29) and one without it (n=31). <b>As an equivalence study the investigators expected that the two techniques were equivalent.</b> Statistics: Descriptive statistics for global description. Student's t test for quantitative variables and chi square test for qualitative variables. Considering statistically significant a p-value less than 0.05. <b>Being an equivalence study, the default delta generated by the Stata command "equim" was used to demonstrate the equivalence between both groups.</b> Results: Demographic data and diagnosis were comparable in both groups (p=NS). No anastomotic leakage or entero-cutaneous fistulae was found in any patient. The investigators demonstrated equivalency since each confidence interval is entirely contained within delta, except for one variable (beginning deambulation), in which equivalency is suggested. There were no significant differences between groups in abdominal distention, infection, or hospital stay variables. Only one patient in the experimental group required placement of the nasogastric tube due to persistent abdominal distension (3.2%). Conclusions. The routine use of nasogastric drainage can be eliminated after distal elective intestinal surgery in children. It's use should be individualized.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 1 month to 18 years old that required elective laparotomy with an intestinal anastomosis (jejunum, ileum and colon).

Exclusion Criteria:

* Non elective anastomosis and high risk groups:

  * newborns
  * upper gastrointestinal tract anastomoses (esophagus, gastric, duodenal or jejunal)
  * bilious-digestive or rectal anastomoses
  * immunosuppressed patients
  * gastrostomy or any pre anastomotic derivation
  * multiple anastomoses
  * chronic intestinal obstruction
  * intraoperative fluids-electrolyte disorders
  * reductive enteroplasty (tapering)
  * emergency operations and patients who did not complete the minimum POP follow up of one month.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2000-09; Primary Completion 2001-04 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
beginning peristalsis, beginning bowel movement, beginning ambulation, time to full diet intake, post-operative stay. | first 5 postoperative days

SECONDARY OUTCOMES:
mild and persistent vomiting, persistent abdominal distention, wound infection or dehiscence, gastrointestinal bleeding, and chief complaint as well as anastomotic leak or dehiscence, reoperation and death. | first 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTO DAVILA, SURGEON, Principal Investigator — Hospital Infantil de Mexico Federico Gomez; EDUARDO BRACHO-BLANCHET, SURGEON, Study Chair — HOSPITAL INFATIL DE MEXICO FEDERICO GOMEZ; JOSE MANUEL TOVILLA-MERCADO, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; RICARDO REYES-RETANA, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; PABLO LEZAMA-DEL-VALLE, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; JOSE ALEJANDRO HERNANDEZ-PLATA, SURGERY, Study Chair — HOSPITAL INFANTIL DE MEXICO; FERNANDO MONTES-TAPIA, SURGERY, Study Chair — HOSPITAL INFANTIL DE MEXICO; ALFONSO REYES-LOPEZ, STATISTIC, Study Chair — HOSPITAL INFANTIL DE MEXICO; JAIME NIETO-ZERMEÑO, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO
Locations (1):
- Hospital Infantil de Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Dinsmore JE, Maxson RT, Johnson DD, Jackson RJ, Wagner CW, Smith SD. Is nasogastric tube decompression necessary after major abdominal surgery in children? J Pediatr Surg. 1997 Jul;32(7):982-4; discussion 984-5. doi: 10.1016/s0022-3468(97)90382-1. PMID 9247217
- [Background] Sandler AD, Evans D, Ein SH. To tube or not to tube: do infants and children need post-laparotomy gastric decompression? Pediatr Surg Int. 1998 Jul;13(5-6):411-3. doi: 10.1007/s003830050351. PMID 9639629
- [Background] Argov S, Goldstein I, Barzilai A. Is routine use of the nasogastric tube justified in upper abdominal surgery? Am J Surg. 1980 Jun;139(6):849-50. doi: 10.1016/0002-9610(80)90395-5. PMID 7386740
- [Background] Cheatham ML, Chapman WC, Key SP, Sawyers JL. A meta-analysis of selective versus routine nasogastric decompression after elective laparotomy. Ann Surg. 1995 May;221(5):469-76; discussion 476-8. doi: 10.1097/00000658-199505000-00004. PMID 7748028
- [Background] Wolff BG, Pembeton JH, van Heerden JA, Beart RW Jr, Nivatvongs S, Devine RM, Dozois RR, Ilstrup DM. Elective colon and rectal surgery without nasogastric decompression. A prospective, randomized trial. Ann Surg. 1989 Jun;209(6):670-3; discussion 673-5. doi: 10.1097/00000658-198906000-00003. PMID 2658880
- [Background] Savassi-Rocha PR, Conceicao SA, Ferreira JT, Diniz MT, Campos IC, Fernandes VA, Garavini D, Castro LP. Evaluation of the routine use of the nasogastric tube in digestive operation by a prospective controlled study. Surg Gynecol Obstet. 1992 Apr;174(4):317-20. PMID 1553612
- [Background] Cunningham J, Temple WJ, Langevin JM, Kortbeek J. A prospective randomized trial of routine postoperative nasogastric decompression in patients with bowel anastomosis. Can J Surg. 1992 Dec;35(6):629-32. PMID 1458389
- [Background] Ordorica-Flores RM, Bracho-Blanchet E, Nieto-Zermeno J, Reyes-Retana R, Tovilla-Mercado JM, Leon-Villanueva V, Varela-Fascinetto G. Intestinal anastomosis in children: a comparative study between two different techniques. J Pediatr Surg. 1998 Dec;33(12):1757-9. doi: 10.1016/s0022-3468(98)90279-2. PMID 9869045
- [Background] Nelson R, Tse B, Edwards S. Systematic review of prophylactic nasogastric decompression after abdominal operations. Br J Surg. 2005 Jun;92(6):673-80. doi: 10.1002/bjs.5090. PMID 15912492
- [Background] Nelson R, Edwards S, Tse B. Prophylactic nasogastric decompression after abdominal surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD004929. doi: 10.1002/14651858.CD004929.pub3. PMID 17636780
- [Background] Rogers JL, Howard KI, Vessey JT. Using significance tests to evaluate equivalence between two experimental groups. Psychol Bull. 1993 May;113(3):553-65. doi: 10.1037/0033-2909.113.3.553. PMID 8316613